CLINICAL TRIAL: NCT06158230
Title: Comparison of Efficacy Between Combination of Amitriptyline-propranolol and Pizotifen for Migraine Prophylaxis: A Single-blind Randomized Controlled Trial
Brief Title: Comparison of Efficacy Between Combination of Amitriptyline-propranolol and Pizotifen for Migraine Prophylaxis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Khandakar Rashed Ahmed, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4292
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Pizotyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amitriptyline-Propranolol (Active Comparator): Combination of amitriptyline and propranolol.
  Initial 2 weeks:
  Amitriptyline 10 mg at bedtime Propranolol 20mg twice daily
  Next 2 weeks:
  Amitriptyline 25 mg at bedtime Propranolol 20mg three times daily
  Next 8 weeks:
  Amitriptyline 25 mg at bedtime Propranolol 40mg twice daily
  Interventions: Drug: Amitriptyline-propranolol
- Pizotifen (Experimental): Pizotifen
  Initial 2 weeks:
  Pizotifen 0.5 mg at bedtime
  Next 2 weeks:
  Pizotifen 1 mg at bedtime
  Next 8 weeks:
  Pizotifen 1.5 mg at bedtime
  Interventions: Drug: Pizotifen

INTERVENTIONS:
Drug: Pizotifen — Pizotifen will be given only at night time to avoid daytime somnolence. Starting dose will be 0.5mg then gradually increased to 1.5 mg
  Arms: Pizotifen
Drug: Amitriptyline-propranolol — Amitriptyline will be given at bedtime only, starting at 10 mg daily and gradually increasing to 25 mg daily.
  Propranolol will be started in 40 mg daily in divided doses, which gradually increases to 80 mg daily in divided doses
  Arms: Amitriptyline-Propranolol

SUMMARY:
The goal of this clinical trial is to compare efficacy and observe common adverse effects of a combination of amitriptyline-propranolol and pizotifen as prophylactic treatments for migraine. The main question it aims to answer is:

• Does pizotifen more effective than the combination of amitriptyline-propranolol in migraine prophylaxis?

Participants will be asked to :

* Maintain the provided headache diary accordingly
* Take supplied drugs as described during clinical visits
* Contact principle investigator if there is any issues regarding drug use and/or their adverse effects

ELIGIBILITY:
Inclusion Criteria:

1. Patient of migraine (with typical aura or without aura) according to ICHD-3 (International Classification of Headache Disorder, 3rd edition) criteria.
2. Age at entry: 18 to 50 years (to minimize the risks related to adverse effects of study drugs such as drowsiness, weight gain, A-V conduction block, postural hypotension)
3. Patients not on any prophylactic medications.
4. Patients willing to take part in the study.
5. Patients being able to fill a headache diary successfully & reliably.

Exclusion Criteria:

1. Age <18 years or >50 years
2. Patients having headache other than migraine, complicated migraine, ophthalmoplegic migraine, catamenial migraine, basilar migraine.
3. Patients on prophylactic medication.
4. Co-morbidities such as heart failure, hepatic or renal impairment, diabetes, bronchial asthma, malignancy, intracranial vascular aneurysm, pregnancy & breastfeeding etc.
5. Patients having known hypersensitivity to amitriptyline, propranolol or pizotifen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2023-03-19 (Actual); Primary Completion 2023-11-25 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of headache per month | 12 weeks
  Comparison of reduction of frequency of headache attack in immediate last month with initial baseline one month without any medication. These values will be compared between two study groups
Duration of headache per month | 12 weeks
  Comparison of reduction of total duration of headache attack in immediate last month with initial baseline one month without any medication. These values will be compared between two study groups
Severity of headache | 12 weeks
  Comparison of reduction of severity of headache attack in immediate last month with initial baseline one month without any medication using visual analogue scale. The visual analogue scale is numbered from 0 to 10. 0 stands for no pain, 1-3 for mild pain, 4-6 for moderate pain and 7-9 for severe pain and 10 for very severe unbearable pain. These values will be compared between two study groups

SECONDARY OUTCOMES:
Adverse effects of drugs | 12 weeks
  Adverse effects (e.g., somnolence, dizziness, dry mouth, weight gain, constipation, bradycardia) of study drugs will be observed

CONTACTS AND LOCATIONS:
Overall Officials: Kanuj Kumar, MD, Study Chair — Professor
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April-2024 to March 2025

REFERENCES:
- [Background] Islam MA, Shaikh AK, AlamSkM, Sultana D, Islam MS, Rashid MM. Safety and Efficacy of Propranolol and amitriptyline combination therapy in migraine prophylaxis: A Randomized Control Trial. J NatlInstNeurosci Bangladesh, 2018;4(1): 3-7
- [Background] Israil A, Ahmed S, Rahman KM, Uddin MJ, Dey SK, Battacharjee M, Mondal G, Ali MA, Alam MN, Miah AH, Uddin MS. Efficacy of amitriptyline, pizotifen and propranolol in the prevention of migraine. Mymensingh Med J. 2013 Jan;22(1):93-100. PMID 23416816
- [Background] Chitsaz, A., Najafi, M.R., Zangeneh, F.A., Norouzi, R. and Salari, M., 2012. Pizotifen in migraine prevention: A comparison with sodium valproate. Neurology Asia, 17(4), pp.319-324.